CLINICAL TRIAL: NCT01000012
Title: Compassionate Use of the Becker Expander/Breast Implant
Status: No longer available | Type: Expanded Access
Sponsor: Mentor Worldwide, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: A101-0501-08cu
Record Dates: First submitted 2009-10-21; First posted 2009-10-22 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-10

CONDITIONS: Breast Reconstruction
MeSH Terms: interventions — Breast Implants

INTERVENTIONS:
Device: Becker 50 Expander/Breast implant — The breast implant is comprised of the Becker implant and the injection dome/fill tube and has a low bleed, gel-filled outer lumen and an adjustable saline-fillable inner lumen. The inner lumen can be gradually filled with saline over an extended period of time via the fill tube by injecting saline through the injection dome. Once expanded to the desired volume, the fill tube and injection dome are removed through a small incision under local anesthetic, and the prosthesis remains in position as a breast implant.
  The Becker 50 Expander/Breast Implant has a 50% gel volume and a 50% saline volume, so a 400cc implant would nominally have 200cc of saline and 200cc of silicone. The Becker 50 Expander/Breast Implant is available in sizes from 300 to 700cc.
Device: Becker 25 Expander/Breast implant — The breast implant is comprised of the Becker implant and the injection dome/fill tube and has a low bleed, gel-filled outer lumen and an adjustable saline-fillable inner lumen. The inner lumen can be gradually filled with saline over an extended period of time via the fill tube by injecting saline through the injection dome. Once expanded to the desired volume, the fill tube and injection dome are removed through a small incision under local anesthetic, and the prosthesis remains in position as a breast implant.
  The Becker 25 Expander/Breast Implant has a silicone gel volume of approximately 25% and saline volume of approximately 75%. The Becker Expander/Breast Implant is available in sizes 150 - 800cc.

SUMMARY:
To provide access of the Becker Expander/Breast implant to women who do not meet inclusion/exclusion criteria of the Becker Continued Access Study

Patients' physician will contact Mentor to request use of the device and each request will be reviewed by Mentor, an IRB, and the FDA on a case-by-case basis

ELIGIBILITY:
Inclusion Criteria:

* Women who require a Becker Expander/Breast implant who do not meet inclusion/exclusion criteria of the Becker Continued Access Study

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Mentor Worldwide LLC, Santa Barbara, California, United States